CLINICAL TRIAL: NCT00829439
Title: A Dose-escalation Tolerability Study of Levodopa/Carbidopa in Angelman Syndrome
Brief Title: Study on Tolerability of Levodopa/Carbidopa in Children With Angelman Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Wen-Hann Tan, Attending Physician in Genetics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-10-0490
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-09

CONDITIONS: Angelman Syndrome
Keywords: Angelman syndrome; Levodopa; Carbidopa; L-dopa
MeSH Terms: conditions — Angelman Syndrome | interventions — Levodopa; Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Levodopa/Carbidopa (Experimental): Other Names:
  Sinemet L-dopa
  Dosages are based on levodopa.
  Each cohort of 3 subjects will be placed on an increasing dose of levodopa (2, 5, 10, and 15 mg/kg/day) for 1 week, provided subjects in the preceding cohort tolerated the lower dose.
  Levodopa/Carbidopa is a combined formulation that will be dispensed as capsules. It should be taken 3 times a day.
  Interventions: Drug: Levodopa/Carbidopa (4:1)

INTERVENTIONS:
Drug: Levodopa/Carbidopa (4:1) — Dosages are based on levodopa.
  Each cohort of 3 subjects will be placed on an increasing dose of levodopa (2, 5, 10, and 15 mg/kg/day) for 1 week, provided subjects in the preceding cohort tolerated the lower dose.
  Levodopa/Carbidopa is a combined formulation that will be dispensed as capsules. It should be taken 3 times a day.
  Other Names: Sinemet; L-dopa

SUMMARY:
This study is designed to determine the highest dose of levodopa/carbidopa that can be tolerated without any serious side effects by children with Angelman syndrome.

It has been hypothesized that levodopa may lead to an improvement in the neurodevelopment and abnormal movements (e.g. tremors) in children with Angelman syndrome.

Data from this study will be used to design a phase II trial to determine the efficacy of levodopa in treating children with Angelman syndrome.

DETAILED DESCRIPTION:
Levodopa is a prodrug that "delivers" dopamine to the brain. It is usually given with carbidopa, a peripheral decarboxylase inhibitor, to increase the bioavailability of levodopa. Animal studies have suggested that levodopa can reverse the excess phosphorylation of some enzymes involved in synaptic and neuronal function, including calcium/calmodulin-dependent kinase type 2 (CaMKII).

Recently, it was shown that excess phosphorylation of CaMKII may be responsible for some of the neurological deficits seen in Angelman syndrome. Therefore, it is hypothesized that levodopa may lead to an improvement in the neurodevelopment and abnormal movements (e.g. tremors) in children with Angelman syndrome.

Although many children have used levodopa for a variety of medical conditions over the last 30 years, it has not been approved by the Food and Drug Administration (FDA) for use in children, and it has not been formally studied in children with Angelman syndrome, so we do not know what dose of levodopa is most appropriate for children with Angelman syndrome.

Therefore, the purpose of this study is to find out the highest dose of levodopa that children with Angelman syndrome can tolerate without any serious side effects.

Once we know the dose of levodopa that can be tolerated by children with Angelman syndrome, we will conduct a larger follow-up study to find out whether levodopa will lead to an improvement in their development and tremor.

ELIGIBILITY:
Inclusion Criteria:

* Angelman syndrome, confirmed by molecular testing
* Must be willing to come for research visit on 2 days, exactly 1 week apart

Exclusion Criteria:

* On levodopa, carbidopa, or any dopamine agonists in the 2 weeks prior to participation
* Other medical conditions that may be associated with developmental or cognitive delays
* More than 2 clinical seizures per month
* Used monoamine oxidase (MAO) inhibitors within the last 2 weeks
* Used phenytoin within the last 2 weeks
* Used phenothiazines, butyrophenones, and thioxanthenes within last 2 weeks
* Hypersensitive to levodopa or carbidopa
* Cardiovascular disease or instability
* Respiratory diseases, including asthma, emphysema, chronic cough, and shortness of breath
* Liver disease
* Stomach or intestinal ulcers
* Kidney disease
* Hematological problems, including anemia, leucopenia, and thrombocytopenia
* Used investigational drugs/interventions within the past three months

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Hann Tan, BMBS, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Levodopa/Carbidopa 2 mg/kg/Day: Levodopa at 2 mg/kg/day in 3 divided doses
- Levodopa / Carbidopa 5 mg/kg/Day: Levodopa 5 mg/kg/day in 3 divided doses
- Levodopa / Carbidopa 10 mg/kg/Day: Levodopa 10 mg/kg/day in 3 divided doses
- Levodopa / Carbidopa 15 mg/kg/Day: Levodopa / Carbidopa 15 mg/kg/day in 3 divided doses
Period: Overall Study
Arm/Group | Levodopa/Carbidopa 2 mg/kg/Day | Levodopa / Carbidopa 5 mg/kg/Day | Levodopa / Carbidopa 10 mg/kg/Day | Levodopa / Carbidopa 15 mg/kg/Day
Started | 3 | 3 | 6 | 4
Completed | 3 | 3 | 5 | 4
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Levodopa/Carbidopa: Other Names:
  Sinemet L-dopa
  Dosages are based on levodopa.
  Each cohort of 3 subjects will be placed on an increasing dose of levodopa (2, 5, 10, and 15 mg/kg/day) for 1 week, provided subjects in the preceding cohort tolerated the lower dose.
  Levodopa/Carbidopa is a combined formulation that will be dispensed as capsules. It should be taken 3 times a day.
  Levodopa/Carbidopa (4:1): Dosages are based on levodopa.
  Each cohort of 3 subjects will be placed on an increasing dose of levodopa (2, 5, 10, and 15 mg/kg/day) for 1 week, provided subjects in the preceding cohort tolerated the lower dose.
  Levodopa/Carbidopa is a combined formulation that will be dispensed as capsules. It should be taken 3 times a day.
Arm/Group | Levodopa/Carbidopa
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Dose of Levodopa/Carbidopa That Can be Tolerated (Without Any Dose Limiting Toxicity) by at Least 3 Subjects.
Time Frame: 1 week
Measure: Number; unit: mg/kg/day
Arm/Group | Levodopa/Carbidopa
Number analyzed (Participants) | 15
mg/kg/day | 15

ADVERSE EVENTS:
Arm/Group | Levodopa/Carbidopa
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 5/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levodopa/Carbidopa (N=16)
Shaky or Unsteady on feet (Nervous system disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No